CLINICAL TRIAL: NCT05603260
Title: An Explorative Experimental Study to Assess the Feasibility, Acceptability and Effectiveness of Imagery Intervention Techniques in the Treatment of Auditory Vocal Hallucinations
Brief Title: Imagery Interventions for Auditory Vocal Hallucinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hella Janssen (Other)
Responsible Party: Sponsor-Investigator, Hella Janssen, coordinating investigator, Geestelijke Gezondheidszorg Eindhoven (GGzE)
Organization: Geestelijke Gezondheidszorg Eindhoven (GGzE) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL79610.068.21
Record Dates: First submitted 2022-10-17; First posted 2022-11-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Auditory Hallucination; Hearing Voices When No One is Talking; Psychosis
Keywords: Mental imagery; Imagery Intervention techniques; Auditory vocal hallucinations; Hearing voices
MeSH Terms: conditions — Hallucinations; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Four single case series A-B-A within subject designs
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meta-cognitive imagery rescripting techniques (M-Int) (Other): These techniques are developed to reduce the power of an image by changing how the client responds to an image by shifting attention away from it, or by doing something that reinforces that it is just an image and not "real".
  Interventions: Behavioral: Imagery intervention for voice hearing (meta-cognitive imagery rescripting)
- Imagery rescripting techniques (ImRs) (Other): These techniques are developed to update imagery appraisals, by for example adding a helpful other to the image or by imagining the scene from another perspective.
  Interventions: Behavioral: Imagery intervention for voice hearing (Imagery rescripting)
- Promoting positive imagery de novo (Other): These involve creating a new stand-alone positive imagery to help a client to increase his ability to self-soothe and reduce fear.
  Interventions: Behavioral: Imagery intervention for voice hearing (promoting positive imagery de novo)
- Visuospatial working memory tasks (Other): These tasks are also known as imagery competing tasks (such as Tetris) and are used to directly target imagery using a tax visuospatial working memory task to reduce the frequency of intrusive imagery.
  Interventions: Behavioral: Imagery intervention for voice hearing (visuospatial working memory tasks)

INTERVENTIONS:
Behavioral: Imagery intervention for voice hearing (meta-cognitive imagery rescripting) — The participants receive intervention for a period of 3 weeks, 6 sessions of 60 minutes.
  In-depth identification of images (2 sessions): Identifying imagery which is related to the auditory vocal hallucinations, constructing a micro-formulation with the participant along the lines of regular Cognitive Behavioural Therapy. In this micro-formulation, first triggers of problematic imagery are identified, both quality and appraisals of this image are identified. Subsequent maladaptive behaviour and possible links with earlier experiences are described, as well as maintaining factors.
  Imagery intervention (2 sessions): The imagery intervention consists of meta-cognitive imagery rescripting.
  Consolidation (2 sessions): Relapse prevention strategies are practiced before the end of intervention.
  Arms: Meta-cognitive imagery rescripting techniques (M-Int)
Behavioral: Imagery intervention for voice hearing (Imagery rescripting) — The participants receive intervention for a period of 3 weeks, 6 sessions of 60 minutes.
  In-depth identification of images (2 sessions): Identifying imagery which is related to the auditory vocal hallucinations, constructing a micro-formulation with the participant along the lines of regular Cognitive Behavioural Therapy. In this micro-formulation, first triggers of problematic imagery are identified, both quality and appraisals of this image are identified. Subsequent maladaptive behaviour and possible links with earlier experiences are described, as well as maintaining factors.
  Imagery intervention (2 sessions): The imagery intervention consists of imagery rescripting.
  Consolidation (2 sessions): Relapse prevention strategies are practiced before the end of intervention.
  Arms: Imagery rescripting techniques (ImRs)
Behavioral: Imagery intervention for voice hearing (promoting positive imagery de novo) — The participants receive intervention for a period of 3 weeks, 6 sessions of 60 minutes.
  In-depth identification of images (2 sessions): Identifying imagery which is related to the auditory vocal hallucinations, constructing a micro-formulation with the participant along the lines of regular Cognitive Behavioural Therapy. In this micro-formulation, first triggers of problematic imagery are identified, both quality and appraisals of this image are identified. Subsequent maladaptive behaviour and possible links with earlier experiences are described, as well as maintaining factors.
  Imagery intervention (2 sessions): The imagery intervention consists of promoting positive imagery de novo.
  Consolidation (2 sessions): Relapse prevention strategies are practiced before the end of intervention.
  Arms: Promoting positive imagery de novo
Behavioral: Imagery intervention for voice hearing (visuospatial working memory tasks) — The participants receive intervention for a period of 3 weeks, 6 sessions of 60 minutes.
  In-depth identification of images (2 sessions): Identifying imagery which is related to the auditory vocal hallucinations, constructing a micro-formulation with the participant along the lines of regular Cognitive Behavioural Therapy. In this micro-formulation, first triggers of problematic imagery are identified, both quality and appraisals of this image are identified. Subsequent maladaptive behaviour and possible links with earlier experiences are described, as well as maintaining factors.
  Imagery intervention (2 sessions): The imagery intervention consists of visuospatial working memory tasks.
  Consolidation (2 sessions): Relapse prevention strategies are practiced before the end of intervention.
  Arms: Visuospatial working memory tasks

SUMMARY:
This study explores the feasibility, acceptability, and effectiveness of four imagery intervention techniques (metacognitive imagery intervention, imagery rescripting, promoting positive imagery and competing imagery task) for auditory vocal hallucinations using four single case series with an A-B-A within subject design.

DETAILED DESCRIPTION:
Auditory vocal hallucinations (AVHs) are the most common hallucinations of psychosis and do often occur in several other mental disorders. The effects of current standard psychological therapy (cognitive behavioural therapy; CBT) for auditory vocal hallucinations are limited. Thus, there is a need to improve cognitive behavioural therapy for auditory vocal hallucinations. As for many other mental disorders specific treatments have been improved using interventions targeting mental imagery, and recent studies pointed towards an association between psychotic symptoms and mental imagery, adding imagery intervention to CBT might aid this aim.

The main objective of this study is to assess the feasibility, acceptability, and effectiveness of four imagery intervention techniques (metacognitive imagery intervention, imagery rescripting, promoting positive imagery and competing imagery task) for auditory vocal hallucinations. The investigators are primarily interested in whether these imagery intervention techniques would be associated with a decrease in auditory vocal hallucinations and imagery symptoms. Also, the investigators are interested in whether these imagery intervention techniques would be a feasible and acceptable intervention for patients with a disorder in the transdiagnostic psychosis and suffering from auditory hallucinations. Secondly, the investigators aim to assess the effects on the level of delusions, visual hallucinations and social and occupational functioning. Lastly, the investigators aim to explore the working mechanisms of imagery, affective symptomatology, and auditory vocal hallucinations by three times daily measuring these symptoms for a period of seven weeks.

The investigators hypothesise that 1) all four imagery interventions are associated with a significant decrease in AVHs (e.g., a decline in the level of auditory vocal hallucinations) and imagery characteristics (e.g., decline in imagery frequency, imagery appraisals and imagery quality), whereas no serious adverse side-effects would occur, drop-out rates of therapy are low and patients will give a good qualitative review of therapy. 2) Psychotic symptoms decrease and social and occupational functioning increase after treatment. 3) The severity of emotional imagery is positively associated with the severity AVHs. In addition, the investigators hypothesize that this association may be different for different imagery aspects, with stronger associations between imagery appraisals (i.e., the encapsulated beliefs, and metacognitive beliefs) and the severity of AVHs as compared to other imagery aspects (frequency and quality aspects). And 4) The associations between imagery related factors and the severity of AVHs are mediated by the level of symptoms of anxiety and depression.

The primary outcome variables, the level of auditory vocal hallucinations and imagery characteristics, are calculated using daily measurements during a two-week baseline, during the intervention and after the end of intervention at follow-up at 7 weeks. Most secondary outcome variables are assessed using self-report measures before baseline, and at pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-65
* Experiencing subclinical or clinical psychotic auditory vocal hallucinations as confirmed by a clinician and as indicated by an intensity score of 4 or more on subscale 1.3 (perceptual abnormalities) of the Comprehensive Assessment of At Risk Mental States (CAARMS) or as indicated by a score of 3 or more on item P3 (hallucinatory behavior) of the Positive and Negative Syndrome Scale (PANSS).
* A Diagnostic and Statistical Manual-5 (DSM-5; American Psychiatric Association, 2013) diagnosis in the psychosis spectrum (codes: DSM-5 codes: 297.1; 298.8; 295.40; 295.90; 295.70; 298.8; 298.9) or defined as Ultra High Risk/At Risk Mental State (ARMS or UHR) according to the CAARMS estimated by a clinician.
* Willing to complete daily monitoring throughout the duration of the study.
* Willing to be assigned to a specific imagery intervention.
* Able to attend 3 consecutive weekly session of imagery intervention and during this period 3 online check-ups.
* Able and willing to sign informed consent

Exclusion Criteria:

* Any current or previous neurological disorder or organic brain disease.
* Acute confusional state or delirium not caused by the psychotic disorder.
* Unwillingness to participate
* Intelligence quotient (IQ) < 70 estimated by clinician.
* Current severe substance or alcohol misuse impacting treatment (clinicians assessment).

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline level of auditory vocal hallucinations to follow-up at two weeks after end of therapy. | Measured three times a day during two weeks of baseline, three weeks of intervention and two weeks of follow-up (an average of 7 weeks)
  Participants received a text message on their mobile phone with a link to a questionnaire. Participants were asked to fill out the questionnaire immediately after the alert, or, if impossible, the same day. All questions will be preceded with the following sentence: "since the last questionnaire….". The questions about auditory vocal hallucinations are adapted from the auditory vocal hallucination rating scale (AVHRS-Q)
Change from baseline level of mental imagery characteristics (frequency of imagery, quality of imagery and appraisals of imagery) to follow-up at two weeks after end of therapy. | Measured three times a day during two weeks of baseline, three weeks of intervention and two weeks of follow-up (an average of 7 weeks)
  Participants received a text message on their mobile phone with a link to a questionnaire. Participants were asked to fill out the questionnaire immediately after the alert, or, if impossible, the same day. All questions will be preceded with the following sentence: "since the last questionnaire….". The questions about mental imagery are adapted from the the Dutch Imagery Survey (DimS)
Treatment safety (change from baseline level of auditory verbal hallucinations to follow-up at the end of therapy). | Administered before baseline period of two weeks, immediately after two weeks of baseline, weekly during the intervention of three weeks and immediately after the end of intervention of three weeks
  The investigators consider treatment to be unsafe if the severity of AVHs of more than 50% of the patients is exacerbated. This will be determined on a case-by-case basis. Worsening of the severity of auditory vocal hallucinations is determined by an increase of 25% as measured with the self-report version of the auditory vocal hallucination rating scale (AVHRS-Q).
Number of Participants with serious adverse events | Administered through study completion, an average of 7 weeks.
  The investigators report the total number of (serious) adverse events
Drop-out rate (i.e., number of participants that drop out) | Administered through study completion, an average of 7 weeks.
  The investigators report drop-outs.
Treatment quality | Administered immediately after the end of intervention of three weeks
  A retrospective self-report assessment is used to evaluate treatment quality. This assessment is based on the retrospective self-report assessment used in a study of one of the co-investigators to evaluate quality of imagery cognitive therapy for bipolar disorders. This is a 32-item self-report questionnaire. Answers are rated on a 5-point Likert scale (ranging from 1 to 5, higher scores indicates a better outcome).

SECONDARY OUTCOMES:
Change in level of social and occupational function from baseline to follow-up at the end of intervention. | Administered before baseline period of two weeks, immediately after two weeks of baseline, and immediately after the end of intervention of three weeks
  measured with the Social and Occupational Functioning Scale (SOFAS). The SOFAS is used to assess overall functioning in a single score. This scale ranges from 0 to 100 (higher score indicates a better outcome), is a modified version of the Global Assessment of Functioning (GAF) scale, separating the measures of social and occupations function from the measure of symptoms, and psychological functioning.
The change from baseline (daily) level of delusional/paranoid ideas to follow-up at two weeks after end of therapy. | Measured three times a day during two weeks of baseline, three weeks of intervention and two weeks of follow-up (an average of 7 weeks)
  This is measured with a visual analogue scale (ranging from 0-100, lower score indicates a better outcome) three times a day with the diary item of delusions.
Change from baseline (daily) level of visual hallucinations to follow-up at two weeks after end of therapy. | Measured three times a day during two weeks of baseline, three weeks of intervention and two weeks of follow-up (an average of 7 weeks)
  This is measured with a visual analogue scale (ranging from 0-100, lower score indicates a better outcome) three times a day with the diary item of visual hallucinations.
Change from baseline imagery characteristics to follow-up at the end of therapy. | Administered before baseline period of two weeks, immediately after two weeks of baseline, and immediately after the end of intervention of three weeks
  Measured with the Dutch Imagery Survey (DimS). The DimS starts with an elaborate definition of imagery. Thereafter, participants are asked to recall and describe an example of an image that is typical of the imagery they have experienced over the previous two weeks. Since studies on imagery and psychoses showed that patients with psychosis experience imagery in relation to their psychotic symptoms, the investigators ask participants to recall the imagery they have experienced in conjunction to their voices in the last two weeks. Participants are instructed to recall this image and keep this image in mind while answering the subsequent questions regarding imagery. All items of the DimS are rated on a 9-point Likert scale (ranging from 1-9). The internal consistency of all subscales of the DiMS are good (Cronbachs alpha ranging from 0.71 to 0.87), consistency over time is also good.

OTHER OUTCOMES:
Mediation variable: Change from baseline level of anxiety to follow-up at two weeks after end of therapy. | Measured three times a day during two weeks of baseline, three weeks of intervention and two weeks of follow-up (an average of 7 weeks)
  Measured daily with a visual analogue scale (ranging from 0-100, lower score indicates a better outcome) three times a day with the diary item of anxiety.
Mediation variable: Change from baseline level of depression to follow-up at two weeks after end of therapy. | Measured three times a day during two weeks of baseline, three weeks of intervention and two weeks of follow-up (an average of 7 weeks)
  Measured daily with a visual analogue scale (ranging from 0-100, lower score indicates a better outcome) three times a day with the diary item of depression.
Mediation variable: Change from baseline level of anxiety to follow-up at the end of intervention. | Administered before baseline period of two weeks, immediately after two weeks of baseline, and immediately after the end of intervention of three weeks
  Measured with Beck Anxiety Inventory (BAI). The BAI is a 21-item self-report questionnaire with good psychometric properties used for measuring the severity of anxiety. Answers are rated on a 4-point Likert scale.
Mediation variable: Change from baseline level of depression to follow-up at the end of intervention. | Administered before baseline period of two weeks, immediately after two weeks of baseline, and immediately after the end of intervention of three weeks
  Measured with the Beck Depression Inventory-II (BDI-II). The BDI-II is widely used self-report questionnaire to assess symptoms of depression and the level of depression. The BDI-II consists of 21 items. Good reliability and validity of the BDI-II have been supported by different studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Geestelijke Gezondheidszorg Eindhoven (GGzE), Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The raw data is generated at the research location and is not shared with other researchers working elsewhere. After publication of the results, only data without privacy sensitive information and without study specific codes (fully anonymous), that support the findings are available from GGzE upon reasonable request (both in and outside the European Union). Before sharing this anonymous data, GGzE carefully investigates this request in consideration of the Dutch AVG and UAVG (Dutch Act on Implementation of the General Data Protection Regulation).

REFERENCES:
- [Background] Hales SA, Di Simplicio M, Iyadurai L, Blackwell SE, Young K, Fairburn CG, Geddes JR, Goodwin GM, Holmes EA. Imagery-Focused Cognitive Therapy (ImCT) for Mood Instability and Anxiety in a Small Sample of Patients with Bipolar Disorder: a Pilot Clinical Audit. Behav Cogn Psychother. 2018 Nov;46(6):706-725. doi: 10.1017/S1352465818000334. Epub 2018 Jul 9. PMID 29983124
- [Background] van den Berg KC, Hendrickson AT, Hales SA, Voncken M, Keijsers GPJ. Comparing the effectiveness of imagery focussed cognitive therapy to group psychoeducation for patients with bipolar disorder: A randomised trial. J Affect Disord. 2023 Jan 1;320:691-700. doi: 10.1016/j.jad.2022.09.160. Epub 2022 Oct 5. PMID 36206888
- [Background] Taylor CDJ, Bee PE, Kelly J, Emsley R, Haddock G. iMAgery focused psychological therapy for persecutory delusions in PSychosis (iMAPS): a multiple baseline experimental case series. Behav Cogn Psychother. 2020 Sep;48(5):530-545. doi: 10.1017/S1352465820000168. Epub 2020 Apr 8. PMID 32264985
- [Background] Ison R, Medoro L, Keen N, Kuipers E. The use of rescripting imagery for people with psychosis who hear voices. Behav Cogn Psychother. 2014 Mar;42(2):129-42. doi: 10.1017/S135246581300057X. Epub 2013 Aug 7. PMID 23920004
- [Background] Paulik G, Steel C, Arntz A. Imagery rescripting for the treatment of trauma in voice hearers: a case series. Behav Cogn Psychother. 2019 Nov;47(6):709-725. doi: 10.1017/S1352465819000237. Epub 2019 Apr 12. PMID 30975230
- [Background] van den Berg KC, Voncken M, Hendrickson AT, Houterman S, Keijsers GPJ. Image qualities and mood variability: Evaluating the utility of an imagery survey for bipolar disorder. J Affect Disord. 2020 Jul 1;272:77-83. doi: 10.1016/j.jad.2020.03.098. Epub 2020 Apr 29. PMID 32379623